CLINICAL TRIAL: NCT01129960
Title: A Phase 3, Double Blind, Randomized, Placebo Controlled, Parallel Group, Multicenter Clinical Study of Eslicarbazepine Acetate in Diabetic Neuropathic Pain
Brief Title: Eslicarbazepine Acetate as Therapy in Diabetic Neuropathic Pain
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BIA-2093-307; 2010-019100-23 (EudraCT Number)
Record Dates: First submitted 2010-05-03; First posted 2010-05-25 (Estimated); Results first posted 2014-07-18 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Painful Diabetic Neuropathy
Keywords: Diabetic Neuropathic Pain
MeSH Terms: conditions — Diabetic Neuropathies | interventions — eslicarbazepine acetate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Eslicarbazepine acetate 800 mg once daily (QD) (Experimental)
  Interventions: Drug: Eslicarbazepine acetate (BIA 2-093)
- Eslicarbazepine acetate 1200 mg QD (Experimental)
  Interventions: Drug: Eslicarbazepine acetate (BIA 2-093)
- Eslicarbazepine acetate 1600 mg QD (Experimental)
  Interventions: Drug: Eslicarbazepine acetate (BIA 2-093)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eslicarbazepine acetate (BIA 2-093) — Tablets will be used.
  Other Names: Exalief; Zebinix; BIA 2-093; ESL
  Arms: Eslicarbazepine acetate 1200 mg QD; Eslicarbazepine acetate 1600 mg QD; Eslicarbazepine acetate 800 mg once daily (QD)
Drug: Placebo — Tablets will be used.
  Arms: Placebo

SUMMARY:
The primary objective of this study is to assess the efficacy of Eslicarbazepine acetate (ESL) as therapy in subjects with Diabetic Neuropathic Pain (DNP) over a 15 week treatment phase.

DETAILED DESCRIPTION:
Diabetic neuropathic pain (DNP) is one of the most common complications of diabetes mellitus. It currently affects about 1% of the population but its prevalence is expected to increase in coming years (European Medicines Agency 2007) in step with the increase in diabetes mellitus prevalence, which is expected to affect 220 million people by 2010

The clinical development of ESL to treat neuropathic pain is based on its chemical and pharmacodynamic relationship to sodium channel blockers, including carbamazepine, which is effective for treating some neuropathic pain conditions. Preclinical data supports the theoretical background.

This study will examine the efficacy, safety, tolerability and pharmacokinetics of Eslicarbazepine acetate for the treatment of diabetic neuropathic pain.

ELIGIBILITY:
Inclusion Criteria:

* Male and female outpatients aged 18 years or older. Female subjects are of nonchildbearing potential, defined as surgical sterilization (hysterectomy or bilateral oophorectomy or tubal ligation) or at least 2 years postmenopausal (spontaneous amenorrhea for at least 24 months before Visit 1), or if of childbearing potential, subjects agree to use a medically acceptable nonhormonal method of contraception.
* Diagnosis of Type 1 or Type 2 diabetes mellitus.
* Pain due to bilateral peripheral polyneuropathy caused by Type 1 or Type 2 diabetes mellitus.
* Have stable glycemic control, as assessed by the investigator, and have glycosylated hemoglobin proportion of less or equal than 11% before randomization.
* A mean score between 4.0 and 9.0, inclusive, on the 24 hour average pain intensity assessment and Visit 3 (ie, 5 of 7 days, 6 of 8 days, 7 of 9 days, or 7 of 10 days).
* Compliance with patient diary completion.
* If not used to treat DNP, subjects are permitted to take nonsteroidal anti inflammatory drugs and selective serotonin reuptake inhibitors if they were kept on a stable dose for 1 month prior to Screening and are foreseen to remain stable throughout the study.
* Competent and able to freely give own informed consent.
* Female subjects of childbearing potential, who are not currently breastfeeding, must have a negative serum pregnancy test at Visit 1.

Exclusion Criteria:

* Historical exposure to drugs known to cause neuropathy.
* Significant skin lesions (active infection, ulcer, etc).
* Peripheral vascular disease with a history of amputation, except amputation of toes.
* Known intolerance to ESL or to other carboxamide derivatives (eg, carbamazepine or oxcarbazepine) or frequent or severe allergic reactions with multiple medications.
* Subjects who previously participated in a clinical study with ESL.
* Major psychiatric disorders.
* Serious or unstable disease that could compromise participation cause hospitalization during the study.
* Second or third degree atrioventricular blockade not corrected with a pacemaker or any clinically significant abnormality in the 12 lead electrocardiogram as determined by the investigator.
* Subjects taking the following drug classes and individual drugs are excluded: benzodiazepines (except short half life sleep agents), skeletal muscle relaxants, orally administered steroids, capsaicin, mexiletine, centrally acting analgesics (dextromethorphan, tramadol), opiates, topical lidocaine, anticonvulsants, tricyclic antidepressants, and serotonin norepinephrine reuptake inhibitors. These drugs require a minimum washout period of at least 5 times the half life and should be tapered appropriately using product label instructions as a guide.
* Relevant clinical laboratory abnormality that, in the investigator's opinion, can compromise the subject's safety.
* History of drug abuse or dependence (drug categories defined by DSM IV) within the past year, excluding nicotine and caffeine.
* Subjects who, in the previous 30 days, received treatment with a drug that had not received regulatory approval for any indication at the time of study entry.
* History of recurrent epileptic seizures except febrile seizures.
* History of severe gastroparesis or gastric bypass surgery.
* Neurolytic treatment for DNP.
* Injected anesthetics or steroid use within 30 days of Visit 1.
* Malignancy within past 2 years.
* History of chronic hepatitis B or C within the past 3 months or human immunodeficiency virus infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332 (Actual)
Dates: Start 2010-11; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- BIAL - Portela & Cª, S.A., S. Mamede Do Coronado, S. Mamede Do Coronado, Portugal

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Fifty nine (59) clinical sites in 10 countries
  Study period:
  Date of first admission: 2010.12.06 Date of last visit: 2012.04.24
Groups:
- Esl 1600 mg: Eslicarbazepine acetate (Esl) (BIA 2-093) mg once daily (QD): Tablets will be used.
- Esl 1200 mg; Esl 800 mg: Eslicarbazepine acetate (BIA 2-093) mg QD: Tablets will be used.
Period: Overall Study
Arm/Group | Esl 1600 mg | Esl 1200 mg | Esl 800 mg | Placebo
Started | 84 | 83 | 82 | 83
Safety | 84 | 83 | 83 (One subject was randomized to placebo, but was dispensed in error with an ESL 800 mg kit at DB Visit) | 82
Intent-to-Treat | 84 | 83 | 82 | 83
Per-Protocol | 34 | 52 | 49 | 55
Full Analysis Set (FAS | 71 | 67 | 68 | 71
Completed | 54 | 61 | 56 | 70
Not Completed | 30 | 22 | 26 | 13
Not completed — Withdrawal by Subject | 3 | 0 | 3 | 2
Not completed — Lack of Efficacy | 1 | 1 | 1 | 1
Not completed — Adverse Event | 23 | 16 | 16 | 7
Not completed — Protocol Violation | 1 | 2 | 3 | 0
Not completed — Lost to Follow-up | 0 | 2 | 3 | 3
Not completed — Discontinuation of the study by Sponsor | 0 | 1 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0
Not completed — Pregnancy | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Esl 1600 mg | Esl 1200 mg | Esl 800 mg | Placebo | Total
Number analyzed (Participants) | 84 | 83 | 83 | 82 | 332
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (10.93) | 59.0 (11.38) | 58.0 (13.33) | 59.5 (10.25) | 58.5 (11.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 35 | 37 | 33 | 150
  Male | 39 | 48 | 46 | 49 | 182
Race/Ethnicity, Customized [Number; unit: participants]
  White | 55 | 50 | 55 | 50 | 210
  Black | 2 | 3 | 1 | 2 | 8
  Asian | 26 | 28 | 25 | 24 | 103
  Other | 1 | 2 | 2 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Endpoint in Mean Pain
Description: Study was prematurely halted. The efficacy analysis was restricted to the primary efficacy variable in the interim analysis population. The intended treatment period, starting on the day of the randomization and ending at the efficacy cut-off date (31st October 2011), was the basis for the efficacy analysis; patients with less than 20 days of study medication were excluded from the analysis, except those with early discontinuation. Primary efficacy variable was the difference between the mean values of 7 daily pain scores preceding the efficacy cut-off date (endpoint mean pain score), and before randomization (baseline mean pain score), respectively. The daily pain scores were based on the morning response to the 11-point Numeric Rating Pain Scale (NRPS) question relating to average pain intensity over the last 24 hours. The NPRS is an 11-point scale from 0-10 ["0" = no pain; "10" = the most intense pain imaginable]
Time Frame: baseline up to endpoint 15 weeks (3-week titration phase and 12-week treatment maintenance phase)
Population: FAS = Full Analysis Set (comprised all randomized subjects with mean pain score at baseline and mean score after randomization; subjects with less than 20 days of study medication of the cut-off date were excluded from the dataset, except those that prematurely withdrew; this was the primary population used in the efficacy analysis)
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Esl 1600 mg | Esl 1200 mg | Esl 800 mg | Placebo
Number analyzed (Participants) | 71 | 67 | 68 | 71
units on a scale | -1.56 (0.232) | -0.90 (0.237) | -1.73 (0.236) | -1.13 (0.231)
Statistical Analysis 1: Comparison: Esl 1600 mg vs Placebo; Test type: Superiority or Other; p = 0.3726, Dunnett's test (analysis of covariance)
Statistical Analysis 2: Comparison: Esl 1200 mg; Test type: Superiority or Other; p = 0.8034, Dunnett's test (analysis of covariance)
Statistical Analysis 3: Comparison: Esl 800 mg vs Placebo; Test type: Superiority or Other; p = 0.1391, Dunnett's test (analysis of covariance)

ADVERSE EVENTS:
Time Frame: Throughout the study
Arm/Group | Esl 1600 mg | Esl 1200 mg | Esl 800 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 5/84 | 3/83 | 1/83 | 6/82
Other Adverse Events (participants affected / at risk) | 53/84 | 38/83 | 35/83 | 10/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Esl 1600 mg (N=84) | Esl 1200 mg (N=83) | Esl 800 mg (N=83) | Placebo (N=82)
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Haemorrhoida haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Diabetic foot infection (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 0
Senile dementia (Nervous system disorders) | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Accelerated hypertension (Vascular disorders) | 1 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Esl 1600 mg (N=84) | Esl 1200 mg (N=83) | Esl 800 mg (N=83) | Placebo (N=82)
Nausea (Gastrointestinal disorders) | 8 | 5 | 10 | 4
Hyponatraemia (Metabolism and nutrition disorders) | 9 | 7 | 2 | 0
Vertigo (Ear and labyrinth disorders) | 9 | 6 | 2 | 0
Somnolence (Nervous system disorders) | 3 | 8 | 4 | 0
Dizziness (Nervous system disorders) | 6 | 3 | 5 | 0
Headache (Nervous system disorders) | 6 | 2 | 6 | 4
Vomiting (Gastrointestinal disorders) | 6 | 3 | 3 | 0
Hypertension (Investigations) | 6 | 4 | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other